CLINICAL TRIAL: NCT01328600
Title: Marinobufagenin as a Target for DIGIBIND in Preeclampsia
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906259; 06-AG-N259
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2014-07-29

CONDITIONS: Preeclampsia
Keywords: Placenta; Pregnancy; Hypertension; Supplementation; Antibody
MeSH Terms: conditions — Pre-Eclampsia; Hypertension

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Preeclampsia is a combination of high blood pressure and other potentially life-threatening symptoms. Preeclampsia occurs in up to 10% of pregnancies and is a main cause of maternal and fetal death worldwide. Treatment is often difficult, and so far there is no specific and effective therapy. Researchers have been studying the body systems that regulate blood pressure. They have also studied drugs that can control certain blood chemicals that constrict blood vessels and increase blood pressure.
* DIGIBIND, a drug that lowers blood pressure, has been used to treat pre-eclampsia. Marinobufagenin (MBG), a chemical in the blood that constricts blood vessels, has been shown to be involved in pre-eclampsia. But researchers are still not certain whether DIGIBIND can be used to specifically target MBG. Researchers want to find out whether DIGIBIND acts against MBG specifically. This information may help them to develop better drugs to block MBG and lower blood pressure in women with preeclampsia.

Objectives:

- To study whether the blood pressure treatment drug DIGIBIND specifically acts on marinobufagenin levels in the blood of pregnant women.

Eligibility:

- Women between 18 and 50 years of age who are 34 to 39 weeks pregnant and have preeclampsia.

Design:

* Participants will be screened with a physical examination, medical history, and blood and urine tests.
* Before delivery, participants will provide blood samples for testing and evaluation.
* Following delivery, participants will provide additional blood samples and samples of the placenta for testing and evaluation.
* No additional treatment, apart from the standard of care, will be provided as part of this protocol.

DETAILED DESCRIPTION:
Preeclampsia (PE) complicates from 5 to 10% of pregnancies and it is a number one cause of maternal and fetal morbidity and mortality worldwide. Nevertheless, a specific and highly effective therapy of this disorder does not exist. As illustrated by therapeutic efficacy of anti-digoxin antibody (DIGIBIND) in preeclampsia, endogenous digitalis-like sodium pump ligands play an important role in the pathogenesis of this syndrome. Previously, we demonstrated that levels of endogenous bufadienolide Na/KATPase inhibitors are elevated in patients with PE, and that antibody to marinobufagenin lower blood pressure in rats with pregnancy-induced hypertension and ex vivo reverse inhibition of the Na/K-ATPase from erythrocytes from patients with PE. Most recently, we developed three anti-MBG monoclonal antibodies which in lower blood pressure in several rat experimental models.

We are proposing a pilot proof-of concept study aimed to demonstrate that MBG is target for DIGIBIND in preeclampsia. If successful, this trial will provide basis for the development of a clinically-usable anti-MBG monoclonal antibody. We hypothesize that in patients with preeclampsia DIGIBIND induces vasorelaxation due to blockade of circulating MBG. The specific aims of the study are to demonstrate that isolated perfused preeclamptic placentae ex vivo release MBG at concentration sufficient to induce vasoconstriction that DIGIBIND reverses vasoconstriction induced by placental perfusate, and that vasorelaxant effect of DIGIBIND is due to blockade of MBG.

The study population will be pregnant women (18-50 years), 34-39 weeks of fetal gestational age with preeclampsia The primary outcome of the study variable will be the difference in the vascular tone in isolated perfused cotyledons. The secondary outcomes will be: (i) the degree of MBG binding to DIGIBIND at different time points following DIGIBIND administration, (ii) the effect of DIGIBIND on the activity of Na/K-ATPase in erythrocytes, and (iii) the ex vivo effect of DIGIBIND on the vascular tone in the isolated placental lobes.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Pregnant women (18-50 years), 34-39 weeks of fetal gestational age with preeclampsia as defined by American College of ObGyn criteria. This definition of PE includes:

   * diastolic blood pressure of at least 90 mm Hg or
   * a systolic blood pressure of at least 140 mm Hg, or
   * a rise in the former of at least 15 mm Hg or in the latter of 30 mm Hg on at least two occasions 6 hours or more apart,
   * proteinuria (presence of 300 mg or more of protein in a 24-hour urine collection or a protein concentration of 1 g or more per liter in at least two random urine specimens collected 6 hours or more apart) or
   * edema (a generalized accumulation of fluid of greater than 1+ pitting edema after 12 hours of bed rest or weight gain of 5 pounds or more in 1 week), or
   * both, induced by pregnancy after the 20th week of gestation, and sometimes earlier.
2. Healthy pregnant women (18-50 years) 34-39 weeks of fetal gestational age as control subjects.
3. Decision of investigator to terminate pregnancy via cesarean section (patient is in need of immediate delivery as soon as clinically appropriate)

EXCLUSION CRITERIA:

1. Eclampsia, i.e., the occurrence of seizures not attributed to another cause during pregnancy
2. Significant antecedent obstetrical problems that may interfere with study assessments or safe participation in the study
3. Evidence of non-reassuring fetal well being
4. Evidence of a lethal or life-threatening fetal anomaly
5. Antecedent hypertension (hypertension secondary to preeclampsia, treated or untreated is allowed)
6. Antecedent renal, hepatic, or autoimmune disease
7. Medical or psychiatric disorders which are unstable or which might interfere with study assessments or safe participation in the study
8. Evidence on medical history/evaluation of use of or need for digitalis-like products currently or in the future
9. Serum creatinine greater than or equal to 1.5 mg/dl
10. Inability to understand and provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2006-08-16; Study Completion 2014-07-29

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Y Bagrov, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (3):
- Russia (3):
  - City Hospital No. 9, Saint Petersburg
  - Pushlon Hospital, Saint Petersburg
  - Veevolozhsk Hospital, Saint Petersburg

REFERENCES:
- [Background] Hamlyn JM, Ringel R, Schaeffer J, Levinson PD, Hamilton BP, Kowarski AA, Blaustein MP. A circulating inhibitor of (Na+ + K+)ATPase associated with essential hypertension. Nature. 1982 Dec 16;300(5893):650-2. doi: 10.1038/300650a0. No abstract available. PMID 6292738
- [Background] Graves SW, Williams GH. An endogenous ouabain-like factor associated with hypertensive pregnant women. J Clin Endocrinol Metab. 1984 Dec;59(6):1070-4. doi: 10.1210/jcem-59-6-1070. PMID 6092405
- [Background] Ludens JH, Clark MA, Kolbasa KP, Hamlyn JM. Digitalis-like factor and ouabain-like compound in plasma of volume-expanded dogs. J Cardiovasc Pharmacol. 1993;22 Suppl 2:S38-41. doi: 10.1097/00005344-199322002-00014. PMID 7508024